CLINICAL TRIAL: NCT05528458
Title: A Phase II Study of Osimertinib to Suppress the Progression of Remaining Ground-glass Opacity Nodule (GGN) for Actionable EGFR Mutation-positive Stage IB-IIIA Lung Adenocarcinoma
Brief Title: Osimertinib to Suppress the Progression of Remaining GGN for EGFR Mutation-positive Stage IB-IIIA Lung Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Se-Hoon Lee, Principle Investigator, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-05-063
Record Dates: First submitted 2022-08-30; First posted 2022-09-06 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Lung Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Osimertinib (Experimental): Subjects should continue on study treatment until objective disease progression, or for three years since osimertinib administration. If progression of remaining GGN on serial CT scan, patients will receive proper treatment for progressed GGN.
  Interventions: Drug: Osimertinib 80Mg Tab
- Obsevation (No Intervention): Subjects with confirmation of pathologic stage IA NSCLC after surgery will be allocated to the control group.

INTERVENTIONS:
Drug: Osimertinib 80Mg Tab — Subjects have a osimertinib (80 mg, orally, once daily) to suppress the progression of remaining GGN(s) in other lobes following surgical resection
  Other Names: Tagrisso
  Arms: Osimertinib

SUMMARY:
This is an open label, phase II study to assess the efficacy of osimertinib (80 mg, orally, once daily) to suppress the progression of remaining GGN(s) in other lobes following surgical resection for actionable EGFR mutation-positive stage IB-IIIA lung adenocarcinoma.

DETAILED DESCRIPTION:
GGN (Ground-glass opacity nodule) is defined as rounded areas of homogeneous or heterogeneous increased attenuation in computed tomography (CT) scans, which are lower in density with regard to surrounding soft tissue structures, such as vessels, that is generally associated with the early-stage lung adenocarcinoma (Lee et al 2011). Therefore, some insist that the malignancy-favored GGO should be called GGN. Multiple pure GGO lesions detected in patients undergoing pulmonary resection for lung adenocarcinoma have a high possibility of malignancy if the size is greater than 7.5 mm. (Kim et al 2009) Nowadays, GGNs of the lung are increasingly detected with thin-section CT scan. GGNs are categorized as pure GGNs and mixed GGNs according to the images from a high-resolution CT.

Usually, lung adenocarcinoma with synchronous GGNs is considered a distinct disease entity in multiple synchronous lung cancers. Few studies have performed next-generation sequencing analysis of these synchronous sequential lesions. Recent study shows that multiple synchronous lesions in the same patient showed different mutation profiles (Park et al 2018) That suggests that adenocarcinoma and synchronous GGNs are genetically independent tumor. But interestingly, driver gene mutations were homogeneously distributed. These findings support the relevance of molecular characterization of lung adenocarcinoma and accompanying GGNs.

The development of a standardized approach to the interpretation and management of GGNs remain critically important given that peripheral adenocarcinomas represent the most common type of lung cancer, with evidence of increasing frequency.

The surgical management of patients with remaining GGN(s) who underwent surgery for the main tumor is still controversial. Although surgical approaches for the remaining lesions depend on their anatomical location, size, and number, as well as the patient's age and pulmonary function, the decision usually depends on the surgeon's judgment; no standard criteria have been established for the selection of the lesions to be treated, nor the method of management of the residual nodules in cases of resectable lung adenocarcinoma with synchronous GGNs. If GGNs are located deep in the hilum or scattered in different lobes or contralateral lung, they cannot be resected simultaneously so that may require additional surgery or radiation therapy. Investiators hypothesized that, in patients with confirmed EGFR mutation positive disease, postoperative osimertinib may regress synchronous GGNs, and eventually, avoid the need of repeated surgery. The purpose of this study is to confirm the efficacy and safety of osimertinib to regress synchronous GGNs in other lobes by osimertinib for stage IB-IIIA adenocarcinoma after curative resection.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Adult male or female patients, aged from 30 to 75 years
3. Pathologic proven lung adenocarcinoma with additional persistent GGNs in at least one other lobe: GGN is defined as a ground glass-opacity with well-defined margin, mean density above -500 HU and greater than 7.5 mm in its maximum diameter
4. The resected lung adenocarcinoma should have actionable EGFR mutation, which is limited to L858R or exon 19 deletion.
5. WHO performance status 0-1 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks
6. Complete surgical resection of the primary NSCLC is mandatory.
7. Uneventful recovery from curative-intent lung cancer surgery

For assignment in the control arm, subjects should be classified post-operatively as Stage IA on the basis of pathologic criteria (the 8th edition of TNM staging system for lung cancer).

For assignment in the treatment arm, subjects should fulfil the following criteria in addition to the above criteria.

* Patients must be classified post-operatively as Stage IB, II or IIIA on the basis of pathologic cirteria (the 8th edition of TNM staging system for lung cancer)
* Female subjects should be using highly effective contraceptive measures, and must have a negative pregnancy test and not be breast-feeding prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

  * Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
  * Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution
  * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation

Further information in Appendix E (Definition of Women of Childbearing Potential and Acceptable Contraceptive Methods)

- Male subjects should be willing to use barrier contraception during the study and for 4 months after last dose of osimertinib

Exclusion Criteria:

1. Regression of synchronous GGN after adjuvant chemotherapy prior to osimertinib
2. Past history of postoperative ALI/ARDS or pneumonia during recovery period
3. Currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of CYP3A4 (at least 3 week prior) (Appendix C). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4.
4. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
5. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib.
6. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 electrocardiograms (ECGs), using the screening clinic ECG machine derived QTc value. Whenever QTc, is mentioned in this document, this refers to correction e made by Fridericia formula (QTcF),
   * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block and second degree heart block.
   * Patient with any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, electrolyte abnormalities (including: Serum/plasma potassium < lower limit of normal (LLN); Serum/plasma magnesium < LLN; Serum/plasma calcium < LLN) , congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval and cause Torsades de Pointes
7. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
8. Inadequate bone marrow reserve or organ function (as demonstrated by any of the following laboratory values:

   * Absolute neutrophil count <1.5 x 109/L;
   * Platelet count <100 x 109/L;
   * Haemoglobin <90 g/L;
   * Alanine aminotransferase >2.5 times upper limit of normal (ULN) if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases;
   * Aspartate aminotransferase >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases;
   * Total bilirubin >1.5 times ULN if no liver metastases or >3 times ULN in the presence of documented Gilbert's Syndrome [unconjugated hyperbilirubinaemia] or liver metastases;
   * Serum creatinine >1.5 times ULN concurrent with creatinine clearance <50 mL/min [measured or calculated by Cockcroft and Gault equation]-confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN.
9. Women who are breast-feeding
10. Males and females of reproductive potential who are not using and effective method of birth control and females who are pregnant or breastfeeding or have a positive (urine or serum) pregnancy test prior to study entry.
11. Involvement in the planning and conduct of the study (applies to AstraZeneca staff or staff at the study site).
12. History of hypersensitivity to active or inactive excipients of osimertinib or drugs with a similar chemical structure or class to osimertinib.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of osimertinib on the regression of additional GGN(s) | The imaging modalities used for GGN assessments will be CT scan (1 mm thin-section) of chest. Baseline, 12weeks, 24weeks, 36weeks, 52weeks and then every 24weeks until 5years assessments should be performed
  Regression rate of each individual GGN using investigator assessments by comparing the size of GGN(s) on the initial CT scan (at screening) to that in the last follow-up scan, assessed by a blinded independent central review (BICR) of the radiologic examination of each patient; We will conduct the quantitative analysis of GGNs on the initial and follow-up CT scans via VOI (Volume of Interest) segmentation. The findings of each GGN on the initial and follow-up CT scans will be analyzed as follows: (1) diameter of the GGO component, (2) diameter of the solid component, (3) volume, (4) mass, (5) density, and (6) a histogram of CT attenuation.
  Regression is defined as follows: (1) disappearance of GGN, 2) more than 25% decrease in longest diameter and no increase of mean density or 3) documented evidence of 25% decrease in kurtosis, skewness, mean density or mass in case of less than 25% decrease in longest diameter

CONTACTS AND LOCATIONS:
Locations (1):
- Sehoon Lee, Seoul, South Korea